CLINICAL TRIAL: NCT03332004
Title: Indocyanine Green and Near-Infrared Vision for Detection of Endometriosis (GRE-Endo Trial)
Brief Title: Near-infrared Fluorescence Imaging as a Supportive Tool for Localisation of Deep Infiltrating Endometriosis During Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GRE-Endo
Record Dates: First submitted 2017-10-12; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Pelvic Endometriosis; Endometriosis Outside Pelvis
Keywords: Indocyanine Green; Deep Infiltrating Endometriosis; Near-Infrared Vision; Occult endometriosis; Invisible endometriosis
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: In the selected patients, after a first white light visual inspection, 0.25 mg/(kg BW) ICG were injected intravenously. After 5 to 30 minutes a second inspection of the abdomen and pelvis in Near Infrared vision was made. All the visualized lesions were carefully described pre and post the Indocyanine Green injection, removed and listed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Indocyanine Green arm (Experimental): All the enrolled patients met the inclusion criteria. No patients have been excluded from the study. All patient have been subjected, during laparoscopy, to an accurate inspection of the abdomen and all the visible endometriotic lesions have been described. Subsequently, 0.25 mg /(kg BW) Indocyanine Green were administered intravenously during surgery and a second look of the abdomen and pelvis with the Near Infrared Vision has been made, in order to identify the fluorescent lesions. All the lesions has been described and localized pre and post the Indocyanine Green injection and then removed and properly cataloged
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — 0.25 mg /(kg BW) Indocyanine Green PULSION® - PULSION Medical Systems were administered intravenously

SUMMARY:
The aim of the study is to establish a new and more accurate method to visualize the peritoneal changes caused by endometriosis using Indocyanine Green mediated fluorescence imaging. The hypothesis is that Indocyanine Green, a fluorescent dye that has wide applications throughout medicine in identifying vascularity of tissues and neovascularization, could facilitate the localization and excision of endometriotic lesions exploiting the hypervascularization due to the chronic inflammation

DETAILED DESCRIPTION:
Patients were recruited within the clinical routine after indication for laparoscopy under consideration of the inclusion and exclusion criteria.

The first abdominal and pelvi's inspection was made using direct laparoscope visualization under white light conditions. All areas suspected of peritoneal endometriosis were classified as white, black and red lesions and recorded together with their anatomic location in the surgical record for the purposes of subsequent extirpation.

After the first visual inspection the patient was administered with 0.05 - 0.25 mg /(kg BW) Indocyanine Green intravenously. The Indocyanine Green imaging mode of the Olympus Indocyanine Green Imaging System was activated and suspected areas in Indocyanine Green imaging mode were recorded with their corresponding appearance in white light mode.

If suspected areas were visible either in white light or Indocyanine Green imaging mode, specific sample has been taken from these areas.

In addition control biopsy specimens from inconspicuous peritoneum has been taken.

ELIGIBILITY:
Inclusion Criteria:

* Suspected endometriosis with necessity for laparoscopic confirmation and resection
* Regular menstrual cycles

Exclusion Criteria:

* Patients younger than 18 years and older than 50 years at time of operation
* Subject with previous history of adverse reaction or allergy to Indocyanine Green, iodine, shellfish or iodine dyes
* Documented allergy to sulfur containing compounds
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Indocyanine Green
* Subject has significant liver disease, cirrhosis or liver insufficiency with abnormal liver function tests (Total bilirubin increased by factor 1.5 than normal and/or serum glutamic oxaloacetic transaminase increased by factor 2 than normal)
* Subject has uremia, serum creatinine (> 2.0 mg/dl)
* Subject has severe coronary heart disease (instable angina pectoris)
* Pregnant or breast-feeding women
* Subject actively participating in another drug, biologic and/or device protocol
* The presence of medical conditions contraindicating general anesthesia or standard surgical approaches
* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-02-16 (Actual)

PRIMARY OUTCOMES:
Detection of endometriotic lesions | Intraoperative
  Optical qualitative assessment through the visual evaluation of a single expert surgeon (presence / absence of fluorescence, due to the injection of the Indocyanine Green and the use of the Near Infrared vision, at the level the of suspected endometriotic lesions)

SECONDARY OUTCOMES:
Localization of occult endometriotic lesion | Intraoperative
  To detect occult endometriotic lesions, thanks to the fluorescence of the Indocyanine Green, that would remain otherwise not visible to the surgeon eye
Operatory Time | Intraoperative
  To assess if the use of Indocyanine Green cause a significant increase of the operatory time
Complications | From operatory room up to 3 days
  To assess if the use of Indocyanine Green increase the percentage of intra and post-operative complications
Side effects | From operatory room up to 3 days
  Evaluation of possible side effects related to the use of Indocyanine Green as a fluorescent endometriosis' marker

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, Principal Investigator — Division of Oncologic Gynecology, Fondazione Policlinico Gemelli
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2013-01-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT03332004/Prot_000.pdf
  • Statistical Analysis Plan (2013-01-29): https://cdn.clinicaltrials.gov/large-docs/04/NCT03332004/SAP_001.pdf